CLINICAL TRIAL: NCT05508789
Title: Global Study to Investigate Safety and Efficacy of Donanemab in Early Symptomatic Alzheimer's Disease
Brief Title: A Study of Donanemab (LY3002813) in Participants With Early Symptomatic Alzheimer's Disease (TRAILBLAZER-ALZ 5)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18442; I5T-MC-AACO (Other: Eli Lilly and Company); 2025-522340-40-00 (EU CTIS Number)
Record Dates: First submitted 2022-08-18; First posted 2022-08-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders
Keywords: Alzheimer's; Dementia; Cognitive Impairment; Amyloid Plaque
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders; Cognitive Dysfunction; Plaque, Amyloid | interventions — donanemab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Donanemab (Experimental): Participants will receive donanemab intravenously (IV)
  Interventions: Drug: Donanemab
- Placebo (Placebo Comparator): Participants will receive placebo IV
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donanemab — Administered IV
  Other Names: (LY3002813)
  Arms: Donanemab
Drug: Placebo — Administered IV
  Arms: Placebo

SUMMARY:
The reason for this study is to assess the safety and efficacy of donanemab in participants with early Alzheimer's disease. The study duration including screening and follow-up is up to 93 weeks.

DETAILED DESCRIPTION:
TRAILBLAZER-ALZ 5 is a Phase 3, double-blind, placebo-controlled study to evaluate the safety and efficacy of donanemab in participants with early symptomatic AD (prodromal AD and mild dementia due to AD) and the presence of AD pathology.

ELIGIBILITY:
Inclusion Criteria:

* Gradual and progressive change in memory function reported by the participant or informant for ≥6 months.
* A MMSE score of 20 to 28 (inclusive) at screening visit.
* Meet amyloid scan (central read) criteria.
* Have a study partner who will provide written informed consent to participate, is in frequent contact with the participant (defined as at least 10 hours per week), and will accompany the participant to the study or be available by telephone at designated times.
* A second study partner may serve as backup. The study partner(s) is/are required to accompany the participant for signing consent. The study partner must be present on all days the cognitive and functional scales are administered.
* If a participant has a second study partner, it is preferred that 1 study partner be primarily responsible for the CDR and the ADCS-ADL assessments.
* Days requiring the following assessments and scales must have a study partner available by telephone if not accompanying participant for the following assessments

  * AEs and concomitant medications
  * CDR, and
  * ADCS-ADL
* Stable concomitant symptomatic AD medications and other medications that may impact cognition for at least approximately 30 days prior to randomization.

Exclusion Criteria:

* Has significant neurological disease affecting the central nervous system other than AD, that may affect cognition or ability to complete the study, including but not limited to, other dementias, serious infection of the brain, Parkinson's disease, multiple concussions, or epilepsy or recurrent seizures (except febrile childhood seizures).
* Has current serious or unstable illnesses including cardiovascular, hepatic, renal, gastroenterologic, respiratory, endocrinologic, neurologic (other than AD), psychiatric, immunologic, or hematologic disease and other conditions that, in the investigator's opinion, could interfere with the analyses in this study; or has a life expectancy of <24 months.
* History of cancer within the last 5 years, except of non-metastatic basal and/or squamous cell carcinoma of the skin, in situ cervical cancer, nonprogressive prostate cancer, or other cancers with low risk of recurrence or spread.
* Contraindication to MRI or PET scans.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline on the Integrated Alzheimer's Disease Rating Scale (iADRS) | Baseline, Week 76
  Change from Baseline on the iADRS in at least one of the low-medium tau pathology population or no-very low and low-medium tau pathology population.

SECONDARY OUTCOMES:
Change from Baseline on the iADRS | Baseline, Week 76
  Change from baseline on the iADRS in the overall population.
Change from Baseline on the Clinical Dementia Rating Scale-Sum of Boxes (CDR-SB) | Baseline, Week 76
  Change from Baseline CDR-SB in at least one of the low-medium tau pathology population, no-very low and low-medium tau pathology populations, and the overall population.
Change from Baseline on the Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog13) Score | Baseline, Week 76
  Change from Baseline on the ADAS-Cog13 Score in the low-medium tau pathology population, no-very low and low-medium tau pathology populations, and the overall population.
Change from Baseline on the Alzheimer's Disease Cooperative Study - instrumental Activities of Daily Living (ADCS-iADL) Score | Baseline, Week 76
  Change from Baseline ADCS-iADL Score in the low-medium tau pathology population, no-very low and low-medium tau pathology populations, and the overall population.
Change from Baseline on the Mini Mental State Examination (MMSE) Score | Baseline, Week 76
  Change from Baseline on the MMSE Score in the low-medium tau pathology population, no-very low and low-medium tau pathology populations, and the overall population.
Change from Baseline in Amyloid Plaque Deposition as by Amyloid Positron Emission Tomography (PET) Scan | Baseline, Week 76
  Change in brain amyloid plaque deposition in the overall population.
Pharmacokinetics (PK): Trough Serum Concentration of Donanemab | Baseline to Week 76
Number of Participants with Treatment-Emergent Anti-Drug Antibodies (ADAs) | Week 76

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (141):
- Argentina (16):
  - Hospital Italiano de Buenos Aires, ABB
  - Clinica Privada Banfield, Banfield
  - Fundación para el Estudio y Tratamiento de Enfermedades Mentales (FETEM), Buenos Aires
  - Stat Research S.A., Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - CIPREC, Buenos Aires
  - Mautalen Salud e Investigación, Buenos Aires
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires
  - Centro Médico Arsema, Buenos Aires
  - Instituto Geriatrico Nuestra Señora de Las Nieves, Buenos Aires
  - Fundación para la Lucha contra las Enfermedades Neurológicas de la Infancia (FLENI), Buenos Aires
  - Centro de Educación Médica e Investigaciones clínicas "Dr. Norberto Quirno" (CEMIC), Buenos Aires
  - IDIM - Instituto de Investigaciones Metabólicas, Ciudad de Buenos Aires
  - INSA Instituto de Neurociencia San Agustin, La Plata
  - Instituto De Investigaciones Clinicas Quilmes, Quilmes
  - INECO Neurociencias Oroño, Rosario
- Australia (16):
  - Emeritus Research, Botany
  - Box Hill Hospital, Box Hill
  - The Prince Charles Hospital, Brisbane
  - NeuroCentrix, Carlton
  - Central Coast Neurosciences Research, Erina
  - Austin Health, Ivanhoe
  - Southern Neurology, Kogarah
  - HammondCare, Malvern
  - The Alfred Hospital, Melbourne
  - Alzheimer's Research Australia, Nedlands
  - The Royal Melbourne Hospital, Parkville
  - St Vincent's Hospital, Sydney
  - KARA Institute for Neurological Diseases, Sydney
  - Central Coast Neurosciences Research (Tumbi Umbi), Tumbi Vmbi
  - Neurodegenerative Disorders Research, West Perth
  - The Queen Elizabeth Hospital, Woodville
- China (50):
  - Beijing Hospital, Beijing
  - Beijing ChaoYang Hospital, Beijing
  - Beijing Friendship Hospital Affiliate of Capital University, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - Beijing Tiantan Hospital Affiliated to Capital Medical University, Beijing
  - Beijing Anding Hospital - Affiliated Capital University of Medical Science, Beijing
  - Beijing Peking Union Medical College Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Xiangya Hospital Central South University, Changsha
  - The Second Xiangya Hospital of Central South University, Changsha
  - Sichuan Provincial People's Hospital, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - The First Afffiliated Hospital of Chongqing Medical University, Chongqing
  - Fujian Medical University Union Hospital-1 Bingfanglou, Fuzhou Fujian
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - Guangzhou First People's Hospital, Guangzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Peking University Sixth Hospital, Haidian District
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Sir Run Run Shaw Hospital, Hangzhou
  - The Second Affiliated hospital of Zhejiang University school of medicine, Hangzhou
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin
  - Jinan Central Hospital, Jinan
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - Nanjing Brain Hospital, Nanjing
  - Shanghai Mental Health Center, Shanghai
  - Shanghai Sixth People's Hospital, Shanghai
  - Huashan Hospital Affiliated Fudan University, Shanghai
  - Shanghai Tongji Hospital, Shanghai
  - Shanghai General Hospital, Shanghai
  - Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai East Hospital, Shanghai
  - The First Hospital of Hebei Medical University, Shijiazhuang
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Huanhu Hospital, Tianjin
  - Tianjin Medical University General Hospital, Tianjin
  - Tongji Hospital Tongji Medical,Science & Technology, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - Wuxi People's Hospital, Wuxi
  - Tangdu Hospital of Fourth Military Medical University of Chinese People's Liberation Army, Xi'an
  - Xianyang Hospital of Yan'an University, Xianyang
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou
  - Xuzhou Central Hospital, Xuzhou
  - Affiliated Hospital of Jiangsu University, Zhenjiang
- Poland (9):
  - Podlaskie Centrum Psychogeriatrii, Bialystok
  - Centrum Medyczne NEUROMED, Bydgoszcz
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk
  - Klinika Neuro-Care, Katowice
  - Diamond Clinic, Krakow
  - Nzoz Neuro-Kard Ilkowski i Partnerzy SPL, Poznan
  - Centrum Medyczne Euromedis, Szczecin
  - Centrum Medyczne NeuroProtect, Warsaw
  - Wroclawskie Centrum Alzheimerowskie, Wroclaw
- South Korea (16):
  - Pusan National University Hospital, Busan
  - Hanyang University Guri Hospital, Guri-si
  - Chonnam National University Hospital, Gwangju
  - Inha University Hospital, Incheon
  - Chungnam national university hospital, Junggu
  - Gachon University Gil Medical Center, Namdong-gu
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Bundang Hospital, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Ewha Womans University Seoul Hospital, Seoul
  - Ajou University Hospital, Suwon
- Spain (8):
  - Barcelonabeta Brain Research Center, Barcelona
  - Fundació ACE, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari de Santa Maria, Lleida
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (11):
  - National Taiwan University Hospital Yun-Lin Branch Dou-Liou Region, Douliu
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao-Sung Dist
  - Cardinal Tien Hospital, New Taipei City
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - New Taipei Municipal TuCheng Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- United Kingdom (15):
  - The Rice Centre - Royal United Hospital, Bath
  - Re:Cognition Health - Birmingham, Birmingham
  - Re:Cognition Health - Bristol, Bristol
  - Surrey and Borders Partnership NHS Foundation Trust, Chertsey
  - Dementia Research Unit, Crowborough
  - Re:Cognition Health - Guildford, Guildford
  - St. George's Hospital, London
  - University College London Hospital, London
  - Re:Cognition Health - London, London
  - Charing Cross Hospital, London
  - Queen's Medical Centre, Nottingham University Hospitals, Nottinghamshire
  - Re:Cognition Health - Plymouth, Plymouth
  - Royal Preston Hospital, Preston
  - Moorgreen Hospital, Southampton
  - Re:Cognition Health - Winchester, Winchester

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Donanemab (LY3002813) in Participants With Early Symptomatic Alzheimer's Disease (TRAILBLAZER-ALZ 5) — https://trials.lilly.com/en-US/trial/356219